CLINICAL TRIAL: NCT02393950
Title: Safety, Tolerability, Pharmacokinetic and Pharmacodynamic Effects of Single Escalating Doses of ODM-106: A Randomised, Double-blind, Placebo-controlled Single Centre Study in Healthy Males
Brief Title: Safety, Tolerability,Pharmacokinetics and Pharmacodynamics of ODM-106 in Healthy Volunteers
Acronym: FIMPAM
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Orion Corporation, Orion Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 3117001; 2014-001317-33 (EudraCT Number)
Record Dates: First submitted 2015-03-06; First posted 2015-03-20 (Estimated); Results first posted 2016-12-23 (Estimated); Last update posted 2016-12-23 (Estimated); Status verified 2016-03

CONDITIONS: Healthy Volunteer Study

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Drug: ODM-106 (Experimental): Oral capsules dosage 2-800mg once daily for one day
  Interventions: Drug: ODM-106
- Drug: Placebo (Placebo Comparator): Oral capsules given once daily for one day
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ODM-106 — Single oral escalating doses of ODM-106 will be administered. Each subject will participate in 4 study periods and will therefore receive 3 single doses of ODM-106 and one single dose of placebo.
  Arms: Drug: ODM-106
Drug: Placebo — Single oral escalating doses of ODM-106 will be administered. Each subject will participate in 4 study periods and will therefore receive 3 single doses of ODM-106 and one single dose of placebo.
  Arms: Drug: Placebo

SUMMARY:
The study is a dose escalation study with 8 planned dose levels. The study is a 4-period crossover design where each healthy volunteer will be randomised to receive three dose levels of ODM-106 (single doses) and one dose of placebo. The study will look at the pharmacokinetics (how the body handles the drug) and pharmacodynamics (how the drug affects the body) of ODM-106.

DETAILED DESCRIPTION:
Eight planned dose levels of ODM-106 will be compared with placebo.There will be 2 panels of subjects with 4 dose levels in each panel. Subjects will be randomised to receive 3 dose levels of active treatment (single doses) and 1 dose of placebo. The dose levels will be escalated from the smallest dose upwards within the study and within the study subject. A third panel of 8 subjects may be included to investigate further dose levels of ODM-106, investigate the effect of taking ODM-106 with food or to compare two different formulations of ODM-106. For an individual subject, the study will consist of a screening period (maximum 4 weeks), 4 study treatment periods with a wash-out period between each study treatment administration and a post-treatment period of about 2 weeks.

The study duration for an individual will be approximately 12-16 weeks. Blood samples will be collected for the assessment of the concentration of ODM-106 and its metabolite.Plasma samples and cumulative urinary samples will be collected for metabolite screening. Safety will be assessed by a 12-lead electrocardiogram (ECG), continuous ECG monitoring, Holter ECG, supine and orthostatic blood pressure and heart rate, body temperature, physical examination, electroencephalogram (EEG), laboratory safety assessments and adverse events. Sedation and psychomotor tests and a quantitative EEG will also be performed.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent obtained.
* Participants must be able to speak, read and understand German.
* Good general health ascertained by detailed medical history and physical examinations.
* Males 18-45 years (inclusive).
* Body mass index (BMI) 18-30 kg/m2 inclusive
* Weight 55-95 kg (inclusive).
* Participants with female partners of child-bearing potential must adhere to a proper form of contraception from first study treatment administration until 3 months after the end-of-study visit.

Exclusion Criteria:

* A predictable poor compliance or inability to understand and comply with protocol requirements, instructions and protocol-stated restrictions or communicate well with the investigator.
* Vulnerable subjects.
* Veins unsuitable for repeated venipuncture.
* Evidence of clinically relevant cardiovascular, renal, hepatic, haematological, gastro-intestinal, pulmonary, metabolic-endocrine, neurological, urogenital or psychiatric disease as judged by the investigator. The participants should be healthy subjects.
* Subjects with a medical history of relevant psychiatric disorders or evidence of significant neuropsychiatric disease
* Any condition requiring regular concomitant medication including herbal products or likely to need any concomitant medication during the study.
* Definite or suspected personal history of hypersensitivity to drugs or excipients.
* Intake of any medication that could affect the outcome of the study, as judged by the investigator, within 2 weeks before first study treatment administration (2 months for enzyme inducing drugs like rifampicin or carbamazepin), or less than 5 times the half-life of the medication.
* A history of alcoholism or excess alcohol intake (including regular consumption of more than 21 units of alcohol per week) .
* Use of nicotine-containing products within 6 months of admission and inability to refrain from using nicotine-containing products during the study.
* History of drug abuse or positive drug screen for amphetamine, barbiturates, benzodiazepines, cannabinoids, cocaine, opiates, methamphetamine or methadone.
* Propensity to get headache when refraining from caffeine-containing beverages.
* Blood donation or loss of clinically relevant amount of blood within 2 months before the screening visit.
* Abnormal 12-lead ECG finding of clinical relevance at the screening visit
* Heart rate (HR) < 50 bpm or > 90 bpm after 10 min in rest (supine) at the screening visit
* At the screening visit: systolic BP < 90 mmHg or > 140 mmHg, diastolic BP < 50 mmHg or > 90 mmHg, orthostatic hypotension decrease of greater than or equal to 20 mmHg for systolic BP, decrease of greater than or equal to 10 mmHg for diastolic BP.
* Abnormal 24-h Holter of clinical relevance at the screening visit,
* Positive serology to human immunodeficiency virus (HIV) antibodies, hepatitis B surface antigen (HBsAg) or hepatitis C virus (HCV) antibodies.
* Any abnormal value of laboratory, vital signs, or physical examination, which may in the opinion of the investigator interfere with the interpretation of the test results or cause a health risk for the subject if he takes part in the study.
* Participation in an investigational drug study within 2 months before entry into this study.
* An employee, a direct or indirect relative of the employee of the contract research organisation or the sponsor.
* Any other condition that in the opinion of the investigator would interfere with the evaluation of the results or constitute a health risk for the subject.
* Subject with abnormal standard EEG judged as clinically relevant by the investigator at screening.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2015-03; Primary Completion 2015-10 (Actual); Study Completion 2016-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rainard Fuhr, MD, Principal Investigator — Parexel International GmbH, Berlin, Germany; John Whiteside, Study Director — Orion Corporation, Orion Pharma
Locations (1):
- Parexel International GmbH, Berlin, Germany

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Healthy male volunteers were recruited
Pre-assignment Details: Screening : Male subjects were screened and following PE, vital signs, EEG, ECG and lab. assessments were randomised into the study.
  Sixteen subjects were randomised to 2 panels of 8, each subject received 3 single doses of ODM-106 and 1 dose of placebo in a randomised crossover design.
  Panel 1 was completed before Panel 2 commenced dosing.
Groups:
- Panel 1: Single oral doses ODM-106 Capsule B: 2, 10, 25, 50 mg , placebo
- Panel 2: Single oral doses ODM-106 Capsule B: 100, 100, 200mg. ODM-106 Capsule A 100 mg , placebo
Period: Overall Study
Arm/Group | Panel 1 | Panel 2
Started | 9 | 9
Period 1 | 8 (6 subjects ODM-106 Capsule B 2 mg and 2 subjects on placebo) | 8 (6 subjects ODM-106 Capsule B 100 mg (1 x 100mg) and 2 subjects on placebo)
Period 2 | 8 (6 subjects ODM-106 Capsule B 10 mg and 2 subjects on placebo) | 8 (6 subjects ODM-106 Capsule B 100 mg (10 x 10mg) and 2 subjects on placebo)
Period 3 | 8 (6 subjects ODM-106 Capsule B 25 mg and 2 subjects on placebo) | 8 (6 subjects ODM-106 Capsule B 200 mg (20 x 10mg) and 2 subjects on placebo)
Period 4 | 8 (6 subjects ODM-106 Capsule B 50 mg and 2 subjects on placebo) | 8 (6 subjects ODM-106 Capsule A 100 mg (10 x 10mg) and 2 subjects on placebo)
Completed | 8 | 8
Not Completed | 1 | 1
Not completed — Adverse Event | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Panel 1: Single oral doses ODM-106 Capsule B 2, 10, 25, 50mg, placebo
- Panel 2: Single oral doses ODM-106 Capsule B 100, 100, 200 mg. ODM-106 Capsule A 100mg, placebo
- Total: Total of all reporting groups
Arm/Group | Panel 1 | Panel 2 | Total
Number analyzed (Participants) | 9 | 9 | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 9 | 9 | 18
  >=65 years | 0 | 0 | 0
Gender [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 9 | 9 | 18
Region of Enrollment [Number; unit: participants]
  Germany | 9 | 9 | 18

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events as a Measure of Safety. Number of Participants With Adverse Events Related to Tolerability.
Description: Clinically relevant changes from baseline in safety laboratory assessments (haematology, clinical chemistry, urinalysis), vital signs (pulse and heart rate), 12 lead electrocardiograms, Holter electrocardiograms, telemetry, physical examination.
Time Frame: From screening up to 16 weeks
Measure: Number; unit: subjects affected
Groups:
- ODM-106 Capsule B 2mg: Single oral dose 2 x 1 mg ODM-106 Capsule B
- ODM-106 Capsule B 10mg: Single oral dose 2 x 5 mg ODM-106 Capsule B
- ODM-106 Capsule B 25mg: Single oral dose 2 x 10mg 1 x 5 mg ODM-106 Capsule B
- ODM-106 Capsule B 50mg: Single oral dose 5 x 10mg ODM-106 Capsule B
- ODM-106 Capsule B 100mg (1 x 100mg): Single oral dose 1 x 100mg ODM-106 Capsule B
- ODM-106 Capsule B 100mg (10 x 10mg): Single oral dose 10 x 10mg ODM-106 Capsule B
- ODM-106 Capsule B 200mg: Single oral dose 20 x 10mg ODM-106 Capsule B
- ODM-106 Capsule A 100mg: Single oral dose 10 x 10mg ODM-106 Capsule A
- Placebo: 2 placebo subjects per Arm with matched number of placebo capsules.
Arm/Group | ODM-106 Capsule B 2mg | ODM-106 Capsule B 10mg | ODM-106 Capsule B 25mg | ODM-106 Capsule B 50mg | ODM-106 Capsule B 100mg (1 x 100mg) | ODM-106 Capsule B 100mg (10 x 10mg) | ODM-106 Capsule B 200mg | ODM-106 Capsule A 100mg | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 16
subjects affected | 0 | 4 | 5 | 1 | 2 | 1 | 3 | 2 | 3

2. Secondary Outcome: Peak Plasma Concentration (cMax) of ODM-106
Description: cMax of ODM-106 after single dosing of either Capsule B or Capsule A
Time Frame: Pre-dose and 15, 30 and 45 min, 1, 1.5, 2, 2.5, 3, 3.5, 4, 6, 8, 12, 24, 48, 72 and 96 hours post dose at each dose level.
Measure: Mean (Standard Deviation); unit: ng/ml
Groups:
- ODM-106 Capsule B 25mg: Single oral dose 2 x 10 mg and 1 x 5 mg ODM-106 Capsule B
- ODM-106 Capsule B 50mg: Single oral dose 5 x 10 mg ODM-106 Capsule B
- ODM-106 Capsule B 100mg (1 x 100mg): Single oral dose 1 x 100 mg ODM-106 Capsule B
- ODM-106 Capsule B 100mg (10 x 10mg): Single oral dose 10 x 10 mg ODM-106 Capsule B
- ODM-106 Capsule B 200mg: Single oral dose 20 x 10 mg ODM-106 Capsule B
- ODM-106 Capsule A 100mg: Single oral dose 10 x 10 mg ODM-106 Capsule A
Arm/Group | ODM-106 Capsule B 2mg | ODM-106 Capsule B 10mg | ODM-106 Capsule B 25mg | ODM-106 Capsule B 50mg | ODM-106 Capsule B 100mg (1 x 100mg) | ODM-106 Capsule B 100mg (10 x 10mg) | ODM-106 Capsule B 200mg | ODM-106 Capsule A 100mg | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 0
ng/ml | 9.1 (4.2) | 18.4 (11.4) | 67.8 (51.7) | 119.2 (60.1) | 22.0 (20.1) | 225.9 (177.2) | 547.7 (319.5) | 8.3 (9.1) |

3. Secondary Outcome: Area Under the Plasma Concentration Versus Time Curve (AUC) of ODM-106
Description: AUC of ODM-106 after single oral dosing of either Capsule B or Capsule A.
Time Frame: Pre-dose and 15, 30 and 45 min, 1, 1.5, 2, 2.5, 3, 3.5, 4, 6, 8, 12, 24, 48, 72 and 96 hours post dose at each dose level. Urine sampling, pre-dose and for 24 hours post dose at each dose level
Measure: Mean (Standard Deviation); unit: h*ng/ml
Arm/Group | ODM-106 Capsule B 2mg | ODM-106 Capsule B 10mg | ODM-106 Capsule B 25mg | ODM-106 Capsule B 50mg | ODM-106 Capsule B 100mg (1 x 100mg) | ODM-106 Capsule B 100mg (10 x 10mg) | ODM-106 Capsule B 200mg | ODM-106 Capsule A 100mg | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 0
h*ng/ml | 16.9 (8.8) | 61.3 (44.1) | 213.8 (78.7) | 559.4 (310.9) | 297.4 (346.3) | 1089.2 (977.0) | 2850.8 (2319.8) | 82.0 (64.7) |

4. Secondary Outcome: Time to Peak Plasma Concentration (Tmax) of ODM-106
Description: tmax of ODM-106 after single oral dosing of Capsule B or Capsule A
Time Frame: as for outcome 2
Measure: Mean (Full Range); unit: h
Groups:
- ODM-106 Capsule B 25mg: Single oral dose 2 x 10 mg 1 x 5mg ODM-106 Capsule B
Arm/Group | ODM-106 Capsule B 2mg | ODM-106 Capsule B 10mg | ODM-106 Capsule B 25mg | ODM-106 Capsule B 50mg | ODM-106 Capsule B 100mg (1 x 100mg) | ODM-106 Capsule B 100mg (10 x 10mg) | ODM-106 Capsule B 200mg | ODM-106 Capsule A 100mg | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 0
h | 0.7 [0.5 to 1.0] | 1.9 [1.5 to 3.0] | 1.5 [0.5 to 3.0] | 2.1 [0.8 to 3.5] | 5.8 [1.5 to 23.9] | 1.5 [0.8 to 3.5] | 1.5 [0.8 to 3.5] | 3.0 [1.5 to 4.0] |

5. Secondary Outcome: Elimination Half-life of ODM-106
Description: Elimination half-life of ODM-106 after single dosing of either Capsule B or Capsule A
Time Frame: as for outcome 2
Measure: Mean (Standard Deviation); unit: h
Groups:
- ODM-106 Capsule B 25mg: Single oral dose 2 x 10 mg 1 x 5 mg ODM-106 Capsule B.
Arm/Group | ODM-106 Capsule B 2mg | ODM-106 Capsule B 10mg | ODM-106 Capsule B 25mg | ODM-106 Capsule B 50mg | ODM-106 Capsule B 100mg (1 x 100mg) | ODM-106 Capsule B 100mg (10 x 10mg) | ODM-106 Capsule B 200mg | ODM-106 Capsule A 100mg | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 0
h | 9.5 (5.5) | 20.6 (12.7) | 23.0 (2.1) | 27.3 (4.7) | 23.5 (6.3) | 27.4 (9.2) | 32.1 (10.0) | 21.7 (3.2) |

6. Secondary Outcome: Metabolite Screening in Plasma and Urine
Description: Metabolite screening in plasma and urine after single dosing
Time Frame: Plasma samples at pre-dose and 15, 30 and 45 min, 1, 1.5, 2, 2.5, 3, 3.5, 4, 6, 8, 12, 24, 48, 72 and 96 hours post dose at each dose level. Urine samples, pre-dose and for 24 hours post dose at each dose level
Reporting Status: Not Posted

7. Secondary Outcome: Effect of ODM-106 on Growth Hormone Levels
Description: Growth hormone levels (Cmax) in serum after single oral dosing with either ODM-106 Capsule B, ODM-106 Capsule A or placebo.
Time Frame: Predose and 1, 2, 3,4, 6 and 8 hours post dose at each dose level.
Population: Only timepoints 2 - 6h evaluated.
Measure: Geometric Mean (Standard Deviation); unit: ng/ml
Arm/Group | ODM-106 Capsule B 2mg | ODM-106 Capsule B 10mg | ODM-106 Capsule B 25mg | ODM-106 Capsule B 50mg | ODM-106 Capsule B 100mg (1 x 100mg) | ODM-106 Capsule B 100mg (10 x 10mg) | ODM-106 Capsule B 200mg | ODM-106 Capsule A 100mg | Placebo
Number analyzed (Participants) | 5 | 5 | 6 | 5 | 6 | 6 | 6 | 6 | 14
ng/ml | 1.7 (3.2) | 0.47 (1.04) | 1.05 (2.88) | 1.93 (1.99) | 0.8 (1.36) | 2.23 (6.12) | 0.82 (0.68) | 4.14 (4.96) | 1.01 (2.45)

8. Secondary Outcome: Sedation Scores on a Visual Analogue Scale (VAS)
Description: Assessment of sedation by subject
Time Frame: Pre-dose and at 1, 6 and 10.5h post dose at each dose level
Reporting Status: Not Posted

9. Secondary Outcome: Dexterity and Reaction Times
Description: Selected battery of psychomotor tests
Time Frame: Pre-dose and at 1 and 6h post dose at each dose level
Reporting Status: Not Posted

10. Secondary Outcome: Quantitative EEG
Description: Quantitative analysis of EEG
Time Frame: Pre-dose and at 1, 6 and 10 h post dose at each dose level
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: From the start of study treatment until the end of study visit (approximately 12-16 weeks)
Description: 16 subjects were randomised into 2 panels of 8 subjects. Each panel of 8 subjects participated in 4 periods as a crossover, during each period 6 subjects received active and 2 subjects received placebo, There was a 2 week washout between each period.
Arm/Group | ODM-106 Capsule B 2mg | ODM-106 Capsule B 10mg | ODM-106 Capsule B 25mg | ODM-106 Capsule B 50mg | ODM-106 Capsule B 100mg (1 x 100mg) | ODM-106 Capsule B 100mg (10 x 10mg) | ODM-106 Capsule B 200mg | ODM-106 Capsule A 100mg | Placebo
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/16
Other Adverse Events (participants affected / at risk) | 0/6 | 4/6 | 5/6 | 1/6 | 2/6 | 1/6 | 3/6 | 2/6 | 3/16
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ODM-106 Capsule B 2mg (N=6) | ODM-106 Capsule B 10mg (N=6) | ODM-106 Capsule B 25mg (N=6) | ODM-106 Capsule B 50mg (N=6) | ODM-106 Capsule B 100mg (1 x 100mg) (N=6) | ODM-106 Capsule B 100mg (10 x 10mg) (N=6) | ODM-106 Capsule B 200mg (N=6) | ODM-106 Capsule A 100mg (N=6) | Placebo (N=16)
SUNBURN (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
RHYTHM IDIOVENTRICULAR (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
VENTRICULAR EXTRASYSTOLES (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
NASAL DRYNESS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PRODUCTIVE COUGH (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
DISTURBANCE IN ATTENTION (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DYSGEUSIA (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
HEADACHE (Nervous system disorders) | 0 (0) | 1 (1) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
EAR DISCOMFORT (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DIARRHOEA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
NAUSEA (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HYPERHIDROSIS (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
RASH (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
MYALGIA (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ABCESS LIMB (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
GASTROENTERITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
NASAL HERPES (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
NASOPHARYNGITIS (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
RHINITIS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
URINARY TRACT INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No